CLINICAL TRIAL: NCT00396578
Title: Aerosolized Antibiotics in Mechanically Ventilated Patients
Brief Title: Aerosolized Antibiotics and Respiratory Tract Infection in Patients on Mechanical Ventilation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Nektar Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORIHS # 2004-3799
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-11

CONDITIONS: Ventilator Associated Pneumonia; Respiratory Infection; Tracheobronchitis
Keywords: aerosolized antibiotics; ventilator associated pneumonia; clinical pulmonary infection score; bacterial resistance
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Respiratory Tract Infections | interventions — Gentamicins

INTERVENTIONS:
Drug: aerosolized vancomycin or gentamicin

SUMMARY:
The purpose of this study was to determine the effect of aerosolized antibiotics on respiratory infection in mechanically ventilated patients.We hypothesize that aerosolized antibiotics , which achieve high drug concentrations in the airway, would more effectively treat respiratory infection, decrease the need for systemic antibiotics and decrease antibiotic resistance.

DETAILED DESCRIPTION:
In patients requiring mechanical ventilation, signs of respiratory infection often persist despite treatment with powerful antibiotics given through the patient's vein. In this trial, patients with purulent secretions were assigned aerosolized antibiotics or placebo by a randomizing protocol. Neither the patients or their doctors knew what the patient was receiving.Need for a systemic antibiotic was determined by the clinical physician. Comparisons were made between placebo and study drug for their effects on pneumonia, respiratory signs of infection, ability to wean patients from the ventilator, systemic(given in the vein) antibiotic use and the development of organisms that were resistant to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* be on mechanical ventilation greater than 3 days
* greater than or equal to 18 years of age survival greater than 14 days
* greater than 2 ccs of tracheal secretions/4 hours

Exclusion Criteria:

* allergy to drugs, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-08; Study Completion 2004-09

PRIMARY OUTCOMES:
Ventilator associated pneumonia Systemic Antibiotic use Clinical pulmonary infection score

SECONDARY OUTCOMES:
Weaning from mechanical ventilation Bacterial resistance

CONTACTS AND LOCATIONS:
Overall Officials: Lucy B Palmer, MD, Principal Investigator — SUNY at Stony Brook
Locations (1):
- University Hospital Medical Center, Stony Brook, New York, United States